CLINICAL TRIAL: NCT02331888
Title: A Prospective, Blinded Clinical Study to Compare the Efficacy Between Three Fetal Monitoring Methods: Electro Uterine Monitor (EUM), Fetal Doppler and Scalp Electrode.
Brief Title: To Compare the Efficacy Between 3 Fetal Monitoring Methods
Acronym: EUM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yariv yogev (Other)
Collaborators: OB-Tools Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Yariv yogev, Prof. Yariv Yogev Director, Division of Obstetrics and Delivery Ward, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0131-14-RMC
Record Dates: First submitted 2014-12-11; First posted 2015-01-06 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Fetal Heartbeat Tracings

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Scalp electrode, fetal doppler and EUM (Experimental): Once in labor, the parturient will be connected to the routine fetal doppler and EUM. When necessary according to clinical indications, the scalp electrode will be connected. Tracing will be recorded simultaneously from all three devices until delivery.
  Interventions: Device: Scalp electrode, fetal doppler and EUM

INTERVENTIONS:
Device: Scalp electrode, fetal doppler and EUM — the parturient will be connected to the routine fetal Doppler and to the EUM. and When necessary to the scalp electrode will be connected. Tracings will be recorded simultaneously from all three devices until delivery. three separate outputs will be processed Output of the scalp electrode recording. Output of the fetal doppler. Output of the EUM. Three noncontinuous segments of 30 minutes each with two segments occurring during the first stage of labor and the third occurring during the second stage of labor, will be randomly picked from the scalp electrode recording with 3 matching segments in time from the EUM100pro and the fetal doppler.

SUMMARY:
Once in labor, the parturient will be connected to the routine fetal doppler and EUM. When necessary according to clinical indications, the scalp electrode will be connected. Tracing will be recorded simultaneously from all three devices until delivery.

DETAILED DESCRIPTION:
Once in labor, the parturient will be connected to the routine fetal doppler and EUM. When necessary according to clinical indications, the scalp electrode will be connected. Tracing will be recorded simultaneously from all three devices until delivery.

study design:

1. signing an informed consent at vas<3
2. admittance to delivery room.
3. Verifying inclusion and exclusion criteria, describing clinical rial goal, motivation and phases.
4. Connecting the patient to three devices (fetal Doppler, scalp electrode and EUM) simultaneously.
5. Recording fetal heart rate until delivery.
6. Disconnecting the patient from all devices if required according to clinical need.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical indication to insert a scalp electrode for fetal heart rate tracing.
2. Maternal age>18 years.
3. Reactive fetal heart rate monitoring and BPP (Biophysical Profile) 8/8 at enrollment.
4. Singleton pregnancy.
5. No fetal abnormality or chromosomal defect.
6. Subjects are willing and able to comply with the requirements of the protocol.
7. Fully understand all elements of, and have singed and dated the written informed consent form before initiation of protocol specified procedures, when vas<3.

Exclusion Criteria:

1. Women who refuse to sign the informed consent form.
2. Maternal age<18 years.
3. Multiple pregnancy.
4. Women with implanted electronic device of any kind.
5. Women with allergic to silver.
6. Irritated skin or open wound.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
The difference between the fetal scalp electrode tracings and the EUM tracings of the fetal heart activity. | 12 month
  Mean Positive Percent Agreement (PPA) for interpretable/un interpretable traces (between EUM, scalp electrode and fetal doppler).

SECONDARY OUTCOMES:
Reliability | 12 months
  Mean sensitivity for individual tracing identification (between EUM, scalp electrode and fetal doppler)
Reliability | 12 months
  Mean Positive Predictive Value (PPV) for individual tracing identification (between EUM, scalp electrode and fetal doppler)
Reliability | 12 months
  The mean False Positive Rate (FPR) for individual tracing identification (between EUM, scalp electrode and fetal Doppler)
Accuracy | 12 months
  The difference in fetal heart rate baseline and variability (between EUM, scalp electrode and fetal doppler)
Accuracy | 12 months
  The difference in periodic changes (between EUM, scalp electrode and fetal Doppler).
Adverse events | 12 months
  Number and percentage of adverse events during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Yariv Yogev, professor, Principal Investigator — Director, division of obstetrics and delivery ward Rabin medical center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel, Israel